CLINICAL TRIAL: NCT04410224
Title: An Open Label, Multicenter, Dose-Finding Clinical Phase 1 Study of ASN004 to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy in Patients With Advanced Malignant Solid Tumors
Brief Title: Study of ASN004 in Patients With Advanced Solid Tumors
Acronym: ASN004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kirilys Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASN004-101
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumor
Keywords: antibody-drug conjugate; immunoconjugate; General Solid Tumors

STUDY DESIGN:
Intervention Model Description: Escalating doses of ASN004
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ASN004 ascending doses (Experimental): Patients will receive escalating doses of ASN004 to identify the best dose for further study.
  Interventions: Drug: ASN004

INTERVENTIONS:
Drug: ASN004 — ASN004 is an antibody-drug conjugate for the treatment of advanced or metastatic solid tumors.

SUMMARY:
Participants in this study will receive ASN004 once every 3 or 4 weeks by intravenous infusion. The ASN004 dosing schedule may be modified based on emerging data and Safety Review Committee decision. The study will test various doses of ASN004 to find out the highest safe dose to test in future trials.

Eligible subjects will be sequentially enrolled in cohorts at escalated doses.

DETAILED DESCRIPTION:
Eligible patients will be sequentially enrolled at escalating doses.

Dose escalation decisions will be based on the review of clinical safety and pharmacokinetic (PD) and pharmacodynamics (PD) data and agreed upon by the Sponsor and investigators.

The maximum tolerated dose (MTD) will have an estimated DLT rate of < 33%. Cohorts may be expanded at any dose level or at the MTD for further evaluation of safety, or PK parameters as required.

ELIGIBILITY:
Inclusion Criteria

1. Provide written, voluntary informed consent prior to any -study specific procedure.
2. Histologically confirmed diagnosis of advanced malignant solid tumor.
3. All patients must agree to provide fresh or archival tumor tissue from the tumor lesion that has not been previously irradiated. Patients without archival tissue may only be enrolled if the patient consents to a screening biopsy and this procedure may be safely performed in the judgment of the Investigator.
4. Evidence of progressive disease.
5. For Dose Expansion patients, eligible tumor histologies will be limited to those malignancies known to have highest expression of 5T4 including colorectal, breast, ovarian, lung, liver, and renal carcinomas. A maximum of 3 prior cytotoxic chemotherapy regimens is permitted for advanced disease.
6. Failure of standard therapy or no standard therapy available.
7. Presence of at least 1 measurable target lesion by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 excluding previously irradiated lesions, bone metastasis, or pleural effusion as sole manifestations of disease. Dose escalation patients with evaluable (non-measurable) disease may be permitted to enroll with Medical Monitor approval.
8. Age of at least 18 years old.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
10. A male patient must agree to use contraception as detailed in this protocol during the treatment period and for at least 3 months after the last dose of study treatment and refrain from donating sperm during this period.
11. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies.

    i. Not a woman of childbearing potential (WOCBP) OR ii. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 3 months after the last dose of study treatment.
12. Adequate organ function.
13. Patients with Mandatory 5T4 Expression: Patients replacing a previously enrolled non-5T4 expressing patient must consent to and provide fresh or archival tumor tissue to the central pathology laboratory for 5T4 immunohistochemistry (IHC) testing. To be eligible, the patient's tumor must be confirmed by the central pathology laboratory to express 5T4 (H score of ≥ 10).
14. Patient is willing and able to comply with all protocol required visits and assessments.

Exclusion Criteria

1. Hematologic malignancies and lymphomas.
2. Patients with known brain metastases unless the patient has a single lesion or multiple lesions whose sum of the longest diameter is ≤ 1 cm AND who are asymptomatic.
3. Serious concurrent medical conditions.
4. Patients with known history of left ventricular ejection fraction of < 50%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of ASN004 | first 21 days for patients administered ASN004 every 3 weeks, and first 28 days for patients administered ASN004 every 4 weeks
  The MTD will be determined by evaluating the number of subjects with treatment related adverse events (AEs) and DLTs.

SECONDARY OUTCOMES:
Calculate the pharmacokinetic (PK) area under the plasma concentration of ASN004 | First 63 days
  Calculate the amount of ASN004 in the bloodstream
Calculate the maximum plasma concentration at steady state | First 63 days
  Calculate the maximum amount of ASN004 in the bloodstream
Calculate the terminal elimination rate of ASN004 | First 63 days
  Calculate how fast ASN004 leaves the body
Change in the size of measurable tumor lesions | up to 1 year
  Change from baseline in the sum of the longest dimension in millimeters or each measurable lesion
Change in the status of non-measurable tumor lesions | Up to 1 year
  Number of subjects that have resolution on non-measurable tumor lesions
Appearance of new tumor lesions | Up to 1 year
  Number of subjects with new lesions

OTHER OUTCOMES:
Correlate 5T4 oncofetal protein (5T4) expression and clinical efficacy | Up to 1 year
  Number of patients with 5T4 expression that have a complete response, partial response or prolonged stable disease when receiving ASN004.

CONTACTS AND LOCATIONS:
Overall Officials: Alison L Hannah, MD, Study Director — Kirilys Therapeutics Inc.
Locations (4):
- United States (4):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - NEXT Oncology, Austin, Texas
  - NEXT Oncology, San Antonio, Texas
  - Next Oncology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No